CLINICAL TRIAL: NCT01226875
Title: Multicentred, Randomized Control Trial Comparing Narrow Versus Wide Focal Zones for Shock Wave Lithotripsy of Renal Calculi
Brief Title: Narrow Versus Wide Focal Zones for Shock Wave Lithotripsy of Renal Calculi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); University of Western Ontario, Canada (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-225
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Kidney Stones
Keywords: SWL; kidney stones; renal calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Narrow focus, LP) (Active Comparator): A (Narrow focus): stone is in lower pole of kidney and SWL using narrow focus on lithotripter
  Interventions: Procedure: SWL: Shock Wave Lithotripsy Intervention
- B (Wide focus, LP) (Active Comparator): B: stone is in lower pole of kidney and SWL using wide focus on lithotripter
  Interventions: Procedure: SWL: Shock Wave Lithotripsy Intervention
- C (Narrow focus, no LP) (Active Comparator): C: stone is in no-lower pole of kidney and SWL using narrow focus on lithotripter
  Interventions: Procedure: SWL: Shock Wave Lithotripsy Intervention
- D (Wide focus, no LP) (Active Comparator): D: stone is in no-lower pole of kidney and SWL using wide focus on lithotripter
  Interventions: Procedure: SWL: Shock Wave Lithotripsy Intervention

INTERVENTIONS:
Procedure: SWL: Shock Wave Lithotripsy Intervention — Shock wave lithotripsy (SWL) is the most common treatment modality for kidney stones. It is a safe and non-invasive treatment performed on patients under intravenous sedation (light anesthesia) on an out-patient basis, whereby shock waves are generated by a source external to the patient's body and are then propagated into the body and focused on a kidney stone. The unique quality of SWL is in its exploitation of shock wave focusing. The Storz lithotripter is an electromagnetic lithotripter with a unique design that allows for a dual focus system with the option of either a narrow (6x28 mm) or wide (9x50 mm) focal zone, depending on the clinical situation. This is the first lithotripter on the market to allow for two different focal zones for shock wave targeting.

SUMMARY:
Shockwave lithotripsy (SWL) is a safe, non-invasive treatment for renal calculi. During SWL energy is focused on in order to break kidney stones and this energy can be varied in size from a narrow (or small) focal zone to a wide (or large) focal zone. This is a multi-centered, randomized study comparing the single treatment success rates of narrow and wide focal zones during SWL.

DETAILED DESCRIPTION:
Shock wave lithotripsy (SWL) is a safe and non-invasive treatment for kidney stones. The SWL machine that is currently in use has a unique feature: the focal zone or the energy that the SWL energy is focused on in order to break kidney stones can be varied in size from a narrow (or small) focal zone to a wide (or large) focal zone. Previous lithotripters have only offered one focal size that corresponded to a narrow range. The objective of this study is to compare the single-treatment success rates of narrow and wide focal zones for the shock wave lithotripsy of renal stones between 5 and 15 mm in greatest diameter, while maintaining a constant overall lithotripsy energy level. A wide focal zone may offer some trade-offs when compared with the traditional narrow focal zone: since the area being treated is larger, it is more likely that the stone will receive adequate energy as it moves with patient breathing during treatment, and less energy per cubic inch will be delivered to the kidney around the stone (which might lead to a lower degree of renal injury); on the other hand less energy per cubic inch will also be delivered to the stone, so that stone fragmentation might be inferior to that with a narrow focal zone. Thus, with this study we want to determine whether there is a significant difference in both stone fragmentation and in renal injury (as measured by the incidence of post-treatment renal hematoma or bruises, and by measuring urinary markers indicating the degree of renal cellular damage). Aside from the random choice of focal zone size, there will be no change to the standard of care for lithotripsy treatment. We predict that the narrow focal shock zone will result in superior stone fragmentation, with higher single-treatment stone free and success rates. However, we may identify a slight increased incidence in the rate of subcapsular renal hematoma and renal damage, as detected by urinary markers.

ELIGIBILITY:
Inclusion Criteria:

* Stone must be radiopaque on a KUB (kidney, ureter and bladder) radiograph, and located within the renal collecting system.
* Patients must have had a CT scan within the past 30 days.
* Stones must be solitary, between 5 and 15 mm in maximal diameter.
* Patient must consent to the trial and be willing to return to their respective lithotripsy unit at 2 weeks and 3 months for follow-up.
* Patients must be treated on the Storz Modulith SLX-F2 machine

Exclusion Criteria:

* More than one renal calculus on the treated side.
* Radiolucent stones (uric acid, indinavir) or cystine stones.
* Stone size < 5 mm and > 15 mm.
* Previous surgical intervention on upper tracts within past five years.
* Congenital anatomic anomalies of the kidney, ureters or bladder (such as calyceal diverticulum, horseshoe kidney, etc.)
* Patient currently taking an α-blocker (alfuzosin, terazosin, doxazosin, tamsulosin, prazosin), calcium channel blocker (verapamil, diltiazem, nifedipine, nicardipine, bepridil, mibefradil), or corticosteroids.
* Pregnancy.
* Age < 18 years.
* Active urinary tract infection.
* Patient exceed weight limit for SWL table (>500 lbs)
* Previous SWL treatment for this stone.
* Uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
SWL efficiency quotient comparison between narrow focus vs wide focus | 2 and 12 weeks
  Comparison of single-treatment lithotripsy success rates at 2 and 12 weeks post-lithotripsy. Successful treatment will be defined as either stone-free status or presence of clinically insignificant asymptomatic residual fragments ≤ 4 mm. SWL efficiency quotient for the treatment groups, as calculated by the standardized formula: % stone-free divided by (100 + % re-treated + % auxiliary procedures).

SECONDARY OUTCOMES:
Incidence of perirenal hematomas | post treatment
  Comparing the narrow and wide foci for the presence of perirenal hematomas post treatment on ultrasound.
Biomarkers for renal injury | day 0; day 1; 1 week
  Comparisons of urinary markers for identifying renal injury
Time to stone passage | 12 weeks
  Time it took to pass the stone for both arms will be compared for the 3 month follow up time.
Pain will be compared between narrow vs wide focus arms | day 0 (post treatment)
  Visual analog pain scores will be compared between arms.
Complication rates | 12 weeks
  Complication rates will be compared between narrow and wide focus treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: John Honey, MD, Principal Investigator — St. Michael's Hospital, University of Toronto; Ken Pace, MD, Principal Investigator — St. Michael's Hospital, University of Toronto; Ben Chew, MD, Principal Investigator — University of British Columbia - Vancouver Coastal Health Research Institute; Ryan Paterson, MD, Principal Investigator — University of British Columbia - Vancouver Coastal Health Research Institute; Hassan Razvi, MD, Principal Investigator — Western University, Canada
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Jim Pattison Pavilion G floor station 5 GI/GU Lithotripsy suite, Vancouver, British Columbia
  - St. Joseph's Hospital, University of Western Ontario, London, Ontario
  - St. Michael's Hospital, University of Toronto, Toronto, Lithotripsy suite, 5th floor Cardinal Carter North Wing, Toronto, Ontario